CLINICAL TRIAL: NCT01089790
Title: A Phase III, Multicenter, Double-blind, Active-Controlled, 52 Week Extension Study to Evaluate the Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus Receiving Background Treatment With Glimepiride Alone or in Combination With Metformin or With Pioglitazone Alone
Brief Title: Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus Receiving Background Treatment With Glimepiride Alone or in Combination With Metformin or With Pioglitazone Alone
Acronym: REDWOOD403
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Phenomix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DUT-MD-403
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dutogliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dutogliptin
- 2 (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Dutogliptin — 400 mg tablet, once daily
  Other Names: PHX1149
  Arms: 1
Drug: Sitagliptin — 100 mg capsule (each capsule contains two 50-mg tablets), once daily
  Other Names: Januvia
  Arms: 2

SUMMARY:
This study will evaluate the long-term safety and efficacy of dutogliptin in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Have successfully completed all required visits of a qualifying Phase 3 core protocol
* Be currently receiving treatment for T2DM as set forth in the qualifying Phase 3 core protocol

Exclusion Criteria:

* Any condition, disease, disorder or clinically relevant laboratory abnormality which, in the opinion of the investigator, would jeopardize the patient's appropriate participation in this study or obscure the effects of treatment

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate safety and tolerability of dutogliptin as assessed by vital signs, adverse event reporting, routine clinical laboratory assessments, and ECG | 52 weeks

SECONDARY OUTCOMES:
To demonstrate maintenance or lowering of HbA1c and fasting plasma glucose. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kaity Posada, PharmD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (149):
- United States (149):
  - Forest Investigative Site 064, Birmingham, Alabama
  - Forest Investigative Site 020, Birmingham, Alabama
  - Forest Investigative Site 025, Muscle Shoals, Alabama
  - Forest Investigative Site 059, Chandler, Arizona
  - Forest Investigative Site 113, Gilbert, Arizona
  - Forest Investigative Site 096, Goodyear, Arizona
  - Forest Investigative Site 080, Peoria, Arizona
  - Forest Investigative Site 098, Phoenix, Arizona
  - Forest Investigative Site 133, Phoenix, Arizona
  - Forest Investigative Site 044, Scottsdale, Arizona
  - Forest Investigative Site 087, Tucson, Arizona
  - Forest Investigative Site 061, Anaheim, California
  - Forest Investigative Site 152, Anaheim, California
  - Forest Investigative Site 041, Chula Vista, California
  - Forest Investigative Site 049, Encinitas, California
  - Forest Investigative Site 022, Greenbrae, California
  - Forest Investigative Site 047, Harbor City, California
  - Forest Investigative Site 010, Huntington Park, California
  - Forest Investigative Site 070, Los Angeles, California
  - Forest Investigative Site 111, Northridge, California
  - Forest Investigative Site 031, Riverside, California
  - Forest Investigative Site 091, Roseville, California
  - Forest Investigative Site 140, Sacramento, California
  - Forest Investigative Site 067, Sacramento, California
  - Forest Investigative Site 145, San Mateo, California
  - Forest Investigative Site 112, Santa Ana, California
  - Forest Investigative Site 128, Tustin, California
  - Forest Investigative Site 011, Walnut Creek, California
  - Forest Investigative Site 063, West Hills, California
  - Forest Investigative Site 115, Colorado Springs, Colorado
  - Forest Investigative Site 088, Denver, Colorado
  - Forest Investigative Site 156, Boca Raton, Florida
  - Forest Investigative Site 148, Brandenton, Florida
  - Forest Investigative Site 073, Clearwater, Florida
  - Forest Investigative Site 004, Daytona Beach, Florida
  - Forest Investigative Site 052, DeLand, Florida
  - Forest Investigative Site 144, Hialeah, Florida
  - Forest Investigative Site 129, Hollywood, Florida
  - Forest Investigative Site 062, Jacksonville, Florida
  - Forest Investigative Site 161, Miami, Florida
  - Forest Investigative Site 157, Miami, Florida
  - Forest Investigative Site 154, Miami, Florida
  - Forest Investigative Site 050, Miami, Florida
  - Forest Investigative Site 122, Miami, Florida
  - Forest Investigative Site 125, Miami Lakes, Florida
  - Forest Investigative Site 069, New Port Richey, Florida
  - Forest Investigative Site 012, Ocala, Florida
  - Forest Investigative Site 015, Orlando, Florida
  - Forest Investigative Site 131, Ormond Beach, Florida
  - Forest Investigative Site 127, Pembroke Pines, Florida
  - Forest Investigative Site 018, Sarasota, Florida
  - Forest Investigative Site 075, St. Petersburg, Florida
  - Forest Investigative Site 138, Tamarac, Florida
  - Forest Investigative Site 026, West Palm Beach, Florida
  - Forest Investigative Site 045, Atlanta, Georgia
  - Forest Investigative Site 079, Augusta, Georgia
  - Forest Investigative Site 077, Decatur, Georgia
  - Forest Investigative Site 042, Dunwoody, Georgia
  - Forest Investigative Site 084, Roswell, Georgia
  - Forest Investigative Site 132, Roswell, Georgia
  - Forest Investigative Site 009, Meridian, Idaho
  - Forest Investigative Site 030, Peoria, Illinois
  - Forest Investigative Site 123, Springfield, Illinois
  - Forest Investigative Site 100, Evansville, Indiana
  - Forest Investigative Site 097, Evansville, Indiana
  - Forest Investigative Site 053, Kansas City, Kansas
  - Forest Investigative Site 008, Wichita, Kansas
  - Forest Investigative Site 078, Erlanger, Kentucky
  - Forest Investigative Site 107, Lexington, Kentucky
  - Forest Investigative Site 024, Madisonville, Kentucky
  - Forest Investigative Site 034, Covington, Louisiana
  - Forest Investigative Site 035, Baltimore, Maryland
  - Forest Investigative Site 046, Oxon Hill, Maryland
  - Forest Investigative Site 165, Rockville, Maryland
  - Forest Investigative Site 003, Brockton, Massachusetts
  - Forest Investigative Site 055, Brockton, Massachusetts
  - Forest Investigative Site 118, New Bedford, Massachusetts
  - Forest Investigative Site 007, Waltham, Massachusetts
  - Forest Investigative Site 163, Cadillac, Michigan
  - Forest Investigative Site 002, Dearborn, Michigan
  - Forest Investigative Site 029, Saint Clair Shores, Michigan
  - Forest Investigative Site 054, Edina, Minnesota
  - Forest Investigative Site 142, St Louis, Missouri
  - Forest Investigative Site 143, St Louis, Missouri
  - Forest Investigative Site 013, Grand Island, Nebraska
  - Forest Investigative Site 150, Omaha, Nebraska
  - Forest Investigative Site 072, Las Vegas, Nevada
  - Forest Investigative Site 065, Las Vegas, Nevada
  - Forest Investigative Site 147, Berkeley Heights, New Jersey
  - Forest Investigative Site 137, Albuquerque, New Mexico
  - Forest Investigative Site 101, Albuquerque, New Mexico
  - Forest Investigative Site 006, Albany, New York
  - Forest Investigative Site 081, New Hyde Park, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 151, New York, New York
  - Forest Investigative Site 155, Asheboro, North Carolina
  - Forest Investigative Site 094, Charlotte, North Carolina
  - Forest Investigative Site 051, Charlotte, North Carolina
  - Forest Investigative Site 117, Charlotte, North Carolina
  - Forest Investigative Site 135, Durham, North Carolina
  - Forest Investigative Site 058, Lenoir, North Carolina
  - Forest Investigative Site 038, Morehead City, North Carolina
  - Forest Investigative Site 040, Salisbury, North Carolina
  - Forest Investigative Site 082, Winston-Salem, North Carolina
  - Forest Investigative Site 039, Akron, Ohio
  - Forest Investigative Site 023, Cincinnati, Ohio
  - Forest Investigative Site 043, Columbus, Ohio
  - Forest Investigative Site 057, Dayton, Ohio
  - Forest Investigative Site 032, Kettering, Ohio
  - Forest Investigative Site 141, Marion, Ohio
  - Forest Investigative Site 159, Marion, Ohio
  - Forest Investigative Site 153, Zanesville, Ohio
  - Forest Investigative Site 083, Bethany, Oklahoma
  - Forest Investigative Site 149, Norman, Oklahoma
  - Forest Investigative Site 102, Ashland, Oregon
  - Forest Investigative Site 005, Eugene, Oregon
  - Forest Investigative Site 001, Medford, Oregon
  - Forest Investigative Site 130, Bensalem, Pennsylvania
  - Forest Investigative Site 037, Harleysville, Pennsylvania
  - Forest Investigative Site 126, Jenkintown, Pennsylvania
  - Forest Investigative Site 158, Morrisville, Pennsylvania
  - Forest Investigative Site 066, Philadelphia, Pennsylvania
  - Forest Investigative Site 036, Tipton, Pennsylvania
  - Forest Investigative Site 103, Greer, South Carolina
  - Forest Investigative Site 090, Manning, South Carolina
  - Forest Investigative Site 033, Pelzer, South Carolina
  - Forest Investigative Site 048, Bristol, Tennessee
  - Forest Investigative Site 114, Chattanooga, Tennessee
  - Forest Investigative Site 104, Chattanooga, Tennessee
  - Forest Investigative Site 099, Arlington, Texas
  - Forest Investigative Site 056, Corpus Christi, Texas
  - Forest Investigative Site 071, Dallas, Texas
  - Forest Investigative Site 017, Dallas, Texas
  - Forest Investigative Site 124, Dallas, Texas
  - Forest Investigative Site 162, DeSoto, Texas
  - Forest Investigative Site 136, Houston, Texas
  - Forest Investigative Site 106, Houston, Texas
  - Forest Investigative Site 014, Irving, Texas
  - Forest Investigative Site 139, Irving, Texas
  - Forest Investigative Site 160, New Braunfels, Texas
  - Forest Investigative Site 146, San Antonio, Texas
  - Forest Investigative Site 109, San Antonio, Texas
  - Forest Investigative Site 119, San Antonio, Texas
  - Forest Investigative Site 076, Salt Lake City, Utah
  - Forest Investigative Site 121, Arlington, Virginia
  - Forest Investigative Site 028, Virginia Beach, Virginia
  - Forest Investigative Site 068, Renton, Washington
  - Forest Investigative Site 092, Spokane, Washington
  - Forest Investigative Site 027, Milwaukee, Wisconsin